CLINICAL TRIAL: NCT02329379
Title: Therapeutic Role of Levothyroxine on the Patients With Atypia of Undetermined Significance (AUS) Goiter
Brief Title: The Role of Levothyroxine on Goiter With Atypia of Undetermined Significance
Acronym: TGAUS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Sheng-Chiang Su (Other)
Responsible Party: Sponsor-Investigator, Sheng-Chiang Su, Attending Physician, National Defense Medical Center, Taiwan
Organization: National Defense Medical Center, Taiwan (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-103-05-081
Record Dates: First submitted 2014-12-29; First posted 2014-12-31 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Goiter
MeSH Terms: conditions — Goiter | interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Unigoiter, ATA (+), AUS (+) on Tx (Experimental): The patients who have uninodular goiter demonstrated by thyroid sono and positive autoantibody of thyroglobulin with pathological reports of fine needle aspiration showing atypical undetermined of significance will take eltroxin for TSH suppression therapy to ameliorate of goiter
  Interventions: Drug: Levothyroxine
- Unigoiter, ATA (-), AUS (+) on Tx (Active Comparator): The patients who have uninodular goiter demonstrated by thyroid sono and negative autoantibody of thyroglobulin with pathological reports of fine needle aspiration showing atypical undetermined of significance will take eltroxin for TSH suppression therapy to ameliorate of goiter
  Interventions: Drug: Levothyroxine
- Unigoiter, ATA (+), AUS (+) without Tx (No Intervention): The patients who have uninodular goiter demonstrated by thyroid sono and positive autoantibody of thyroglobulin with pathological reports of fine needle aspiration showing atypical undetermined of significance decide not to take eltroxin for TSH suppression therapy; instead, only observation with following will be conducted
- Unigoiter, ATA (-), AUS (+) without Tx (No Intervention): The patients who have uninodular goiter demonstrated by thyroid sono and negative autoantibody of thyroglobulin with pathological reports of fine needle aspiration showing atypical undetermined of significance decide not to take eltroxin for TSH suppression therapy; instead, only observation with following will be conducted
- Multigoiter, ATA (+), AUS (+) on Tx (Experimental): The patients who have multinodular goiter demonstrated by thyroid sono and positive autoantibody of thyroglobulin with pathological reports of fine needle aspiration showing atypical undetermined of significance will take eltroxin for TSH suppression therapy to ameliorate of goiter
  Interventions: Drug: Levothyroxine
- Multigoiter, ATA (-), AUS (+) on Tx (Active Comparator): The patients who have multinodular goiter demonstrated by thyroid sono and negative autoantibody of thyroglobulin with pathological reports of fine needle aspiration showing atypical undetermined of significance will take eltroxin for TSH suppression therapy to ameliorate of goiter
  Interventions: Drug: Levothyroxine
- Multigoiter, ATA (+), AUS (+) without Tx (No Intervention): The patients who have multinodular goiter demonstrated by thyroid sono and positive autoantibody of thyroglobulin with pathological reports of fine needle aspiration showing atypical undetermined of significance decide not to take eltroxin for TSH suppression therapy; instead, only observation with following will be conducted
- Multigoiter, ATA (-), AUS (+) without Tx (No Intervention): The patients who have multinodular goiter demonstrated by thyroid sono and negative autoantibody of thyroglobulin with pathological reports of fine needle aspiration showing atypical undetermined of significance decide not to take eltroxin for TSH suppression therapy; instead, only observation with following will be conducted

INTERVENTIONS:
Drug: Levothyroxine
  Other Names: Eltroxin
  Arms: Multigoiter, ATA (+), AUS (+) on Tx; Multigoiter, ATA (-), AUS (+) on Tx; Unigoiter, ATA (+), AUS (+) on Tx; Unigoiter, ATA (-), AUS (+) on Tx

SUMMARY:
1. To elucidate the therapeutic role of levothyroxine on the patient with atypia of undetermined significance (AUS) goiter, we would design a prospective, open label and non-randomized trial to verify the therapeutic effects on goiter with AUS by means of TSH (Thyrotropin; Thyroid-Stimulating Hormone) suppression related reduction of goiter volume with subsequent alleviation of previous cytological malignant tendency. During following for 1-2 years after therapy with simultaneous monitor of possible adverse effects of levothyroxine (eltroxin), we collected blood samples and gathered all necessary data as well as performed thyroid sonography with fine-needle aspiration (FNA) for the subjects. Furthermore, we would finish our individual study for each enrolled subject if his/her condition exhibited the criteria of primary end point: reduced goiter volume under sono >15% or cytology: benign for 2 times; operation for thyroidectomy, CAD attack, refractory arrhythmia, newly DM (Diabetes Mellitus), etc.
2. To re-evaluate the current prevalence of goiter within Taiwanese adults, we recruited all patients who presented possible thyroid related symptoms, such as unexplained body weight loss with increased appetite, palpitation, hand tremors, neck swelling, hoarseness and abnormal sensation over throat. Only the patients with goiter proven by thyroid sono in euthyroid status without other preexisting major disorders can be enrolled in our trial to undergo open label, non-randomized study.

DETAILED DESCRIPTION:
The prevalence of goiter in Taiwanese adults was found to be 19.4% in males, 33.6% in females and 25% in total about 20 years ago even though there was no iodine-deficient area reported in Taiwan. The result implied that goiter not only became a quite common disorder, but also deserved further investigation, particularly since 0.7% of goiter would be diagnosed as thyroid cancers by means of fine-needle aspiration (FNA). However, the recent research indicated 5-15% of results after fine-needle aspiration directly disclosed malignant cytology. On the other hand, about 80% of initial results of FNA would appear non-malignant cytology. The most common feature of them was found to be indeterminate cytology, which refers to 15-30% of FNA specimens. The indeterminate cytology included follicular or Hurthle cell neoplasm as well as atypia of undetermined significance (AUS). Based on the revised American Thyroid Association Management Guidelines for Patients with Thyroid Nodules, people would be referred to visit surgeons for surgical intervention if their reports of FNA demonstrated either Hurthle cell neoplasm or follicular neoplasm without autonomously functioning nodules; instead, population with AUS goiter only received observation for a period of time for following. Otherwise, they would be arranged to undergo surgical manipulations if any evidence of malignancy was suspected. There has been lack of sufficient studies to offer therapeutic options for the patient with AUS goiter around the world up to the present, especially in Taiwan. Therefore, in order to avoid unnecessary operation performed upon the patient with AUS goiter and provide another effective treatment for them, a well-designed, prospective clinical trial will be warranted on the patient with AUS goiter.

To achieve the goal, the pathophysiology of goiter required to be understood at first. Although the actual etiology of goiter was uncertain, TSH (thyrotropin) has been regarded as a major factor to induce its formation up to now. To attenuate the growth-tropic effects of TSH, levothyroxine suppression therapy had been administered in the past to treat goiter, particularly about the goiter with colloid nodules. Successful reduction of goiter volume was found in some published papers while others did not verify the therapeutic effects of levothyroxine. However, the fact that goiter with size under thyroid sonogram more than 1cm required to be further examined indicated reduced volume of goiter may offer benefits including amelioration of previous malignant tendency especially in AUS goiter through TSH suppression therapy though some studies indicated routine suppression therapy of benign thyroid nodules in iodine sufficient populations is not recommended At first, patients who aged 20 to 70 with thyroid dysfunction related manifestations as goiter, palpitation or hand tremors would be recruited while they visited MET OPD (Out-Patient Department) and then they would be arranged to undergo thyroid sono as well as receive thyroid functional tests during screening periods before the study. The patients would be eligible for the interventional trial if their thyroid sonography demonstrated goiter and their thyroidal function revealed euthyroid status. After careful investigations of subjects' associated histories as family histories, drug histories and diet habits, the patients would be actually recruited for the clinical trial with the signed informed consent. Initially, the enrolled subjects would be classified into two major groups as solitary nodular goiter and multiple nodular goiter. Subsequently, two subgroups would be identified from each major group by presence of autoantibody of thyroglobulin or not. Thereafter, the patients would be asked to comply with the guidelines of ATA (American Thyroid Association) for advanced evaluation , fine needle aspiration and following if they indeed present with either goiter with more than 1 cm in size or less than 1 cm with regard to typical malignant characteristics under thyroid sonography, such as heterogeneous, hypoechoic, increased peri-vascularization, tall than wide. Furthermore, patients with history of family MTC (Medullary Thyroid Cancer) or contact of radiation or radiation therapy would be arranged to under FNA, too. The patients with first FNA disclosing AUS (atypia of undetermined significance) would be arranged to receive FNA again for confirmatory examination one month later and soon later those patients with positive findings of AUS twice would be allowed to take eltroxin for TSH suppression therapy. On the contrary, the patients would be assigned to the groups who will receive traditional observation and following of thyroid sonography as well as thyroid functional tests. These observed patients would receive surgical interventions if their FNA showed malignant potentials as NUCLEAR GROOVING， MICROFOLLICULAR FOCI，Hurthle cell, etc.

As to the studied patients with consecutive FNA reports indicating AUS twice would be arranged to take levothyroxine (eltroxin, 0.1 mg) for therapy and its dosage would be adjusted carefully after 2 weeks per each OPD visiting. Optimal therapeutic goals would be regarded as subclinical hyperthyroidism and constant concentrations or dosages of eltroxin would be achieved in 2 months. Thereafter, the studied subjects would be arranged to receive thyroid sonography and FNA 3 months later and other necessary blood biochemistry studies for following. All following information would be recorded well and completely. The primary endpoint means: reduced goiter volume under sono >15% or cytology: benign*2 times; operation for thyroidectomy; CAD attack; refractory arrhythmia; newly DM. The pathology of all FNA during the clinical trial would be judged by the Bethesda System for Reporting Thyroid Cytopathology.

ELIGIBILITY:
Inclusion Criteria:

* all patients who presented with goiter proven by thyroid sono in euthyroid status without other preexisting major disorders and possible thyroid related symptoms, such as unexplained body weight loss with increased appetite, palpitation, hand tremors, neck swelling, hoarseness and abnormal sensation over throat.

Exclusion Criteria:

* all patients without definite goiter
* all patients with major illness as CAD, DM or CVA (CerebroVascular Accident)
* all patients with pregnancy or malignancy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05 (Estimated); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with reduced goiter volume under sono >15% | 2 years
Number of participants with fine-needle aspiration cytology: benign*2 times | 2 years

SECONDARY OUTCOMES:
Number of participants need to receive operation for thyroidectomy due to malignant potentials | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Chiang Su, Principal Investigator — Tri-Service General Hospital National Defense Medical Center